CLINICAL TRIAL: NCT06571942
Title: Effect of the Inhaled Triple Therapies Over the Small Airway in Patients With Chronic Obstructive Pulmonary Disease or Chronic Bronchitis Without Obstruction Secondary to Biomass Exposure: Randomized Controlled Clinical Trial Phase IV
Brief Title: Effect of the Inhaled Triple Therapies Over the Small Airway in Biomass Exposure
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Respiratory Diseases, Mexico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C74-23
Record Dates: First submitted 2024-06-28; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: COPD Bronchitis; Pollution Related Respiratory Disorder
Keywords: Biomass; COPD; Chronic bronchitis; Inhaled therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic | interventions — vilanterol; GSK573719; Beclomethasone; Formoterol Fumarate; Budesonide

STUDY DESIGN:
Intervention Model Description: Study comparing the effect of 3 inhaled triple therapies and 1 inhaled double therapy in small airway in COPD and pre-COPD patients for three months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- COPD due to biomass exposure (Experimental): Vilanterol / Umeclidinium 25/62.5 mcg once daily for three months = ANORO® Fluthicasone / Vilanterol / Umeclidinium 100/25/62.5 mcg once daily for three months = TRELEGY® Beclomethasone / Formoterol / Glycopyrronyum 100/6/12.5 mcg; two inhalations twice daily for three months = TRIMBOW® Budesonide / Formoterol / Glycopyrronyum 160/4.8/7.2 mcg; two inhalations twice daily for three months= TRIXEO®
  Interventions: Drug: Vilanterol / Umeclidinium (25/62.5 mcg); Drug: Fluthicasone / Vilanterol / Umeclidinium (100/25/62.5 mcg); Drug: Beclomethasone / Formoterol / Glycopyrronyum 100/6/12.5 mcg; Drug: Budesonide / Formoterol / Glycopyrronyum 160/4.8/7.2 mcg
- Chronic bronchitis without obstruction due to biomass exposure (Experimental): Vilanterol / Umeclidinium 25/62.5 mcg once daily for three months = ANORO® Fluthicasone / Vilanterol / Umeclidinium 100/25/62.5 mcg once daily for three months = TRELEGY® Beclomethasone / Formoterol / Glycopyrronyum 100/6/12.5 mcg; two inhalations twice daily for three months = TRIMBOW® Budesonide / Formoterol / Glycopyrronyum 160/4.8/7.2 mcg; two inhalations twice daily for three months= TRIXEO®
  Interventions: Drug: Vilanterol / Umeclidinium (25/62.5 mcg); Drug: Fluthicasone / Vilanterol / Umeclidinium (100/25/62.5 mcg); Drug: Beclomethasone / Formoterol / Glycopyrronyum 100/6/12.5 mcg; Drug: Budesonide / Formoterol / Glycopyrronyum 160/4.8/7.2 mcg

INTERVENTIONS:
Drug: Vilanterol / Umeclidinium (25/62.5 mcg) — One inhalation daily from Ellipta device for three months
  Other Names: ANORO
Drug: Fluthicasone / Vilanterol / Umeclidinium (100/25/62.5 mcg) — One inhalation daily from Ellipta device for three months
  Other Names: TRELEGY
Drug: Beclomethasone / Formoterol / Glycopyrronyum 100/6/12.5 mcg — Two inhalations twice daily form pMDI device for three months
  Other Names: TRIMBOW
Drug: Budesonide / Formoterol / Glycopyrronyum 160/4.8/7.2 mcg — Two inhalations twice daily form pMDI device for three months
  Other Names: TRIXEO

SUMMARY:
This phase IV randomized controlled clinical trial intend to compare the effect of three close standard inhaled triple therapies and one close standard inhaled double therapy on the small airway in patients with Chronic Obstructive Pulmonary Disease (COPD-B) and chronic bronchitis without obstruction (BCNO) exposed to wood smoke. The treatment phase duration is of 3 months. As primary outcome, the resistance change in post-bronchodilatator impulse oscilometry will me measure at 30 minutes, 2 hours, 4 hours, and 24 hours post first dose of the asigned medication, and then at 1 and 3 months of treatment. As secondary outcomes, change in respiratory symptoms and health related quality of life will be assess after 1 and 3 months of treatment.

DETAILED DESCRIPTION:
Selection visit day -21 to -1: The diagnosis of COPD-B or BCNO will be verified. The inclusion criteria will be checked and it will be verified if there are any exclusion criteria (clinical record will be reviewed if necessary). The patient is invited to the study, will be given detailed information about it, and a copy of the informed consent for evaluation. If they agree to participate in the study, they will be asked to sign the consent in the indicated space, as well as two witnesses. If the patient does not have post-bronchodilator forced spirometry and a six-minute walk in the last 3 weeks, these tests will be performed in the COPD lung function laboratory. A symptom diary will be dispensed and training will be given on how to fill it out. The patient will be instructed to begin the washout time, which will be one week for long-acting bronchodilators (LAMA or LABA, or LAMA/LABA combination), and 3 weeks for inhaled steroids (or ICS/LABA, ICS/LAMA/LABA). During this period, patients will be able to use their rescue bronchodilator (SAMA, SABA, or combination) by schedule. They will be instructed in the identification of exacerbations and alarm symptoms and, if necessary, communicate with the principal investigator.

Randomization visit and initiation of treatment. (Visit 0, day 0): A complete patient history will be taken, with main emphasis on the recording of comorbidities and concomitant medication. Inclusion and exclusion criteria will be checked. The washout time of each bronchodilator will be confirmed, and once confirmed, baseline questionnaires will be performed: Measurement of dyspnea (mMRC scale) and health realated quality of life questionnaires (CAT and SGRQ). The history of exacerbations in the last 4 weeks will be verified. If the patient continue to meet the criteria, they will be selected and baseline respiratory function tests will begin: The tests will be performed between 7:00 to 8:00 AM in the following order: Exhaled fraction of nitric oxide (FeNO), impulse oscillometry, slow spirometry, forced spirometry, and simple plethysmography. The selection criteria will be confirmed and if they are a candidate, randomization will be carried out through the Redcap program. Patients will be assigned one of the four devices contemplated for the study. The first group will be assigned the device containing Vilanterol/Umeclidinium 25/62.5 mcg (Anoro) with a dose of one inhalation every 24 hours; the second group will be assigned the device containing Fluticasone/ Vilanterol/ Umeclidinium 100/25/62.5 mcg (Trelegy) with a dose of one inhalation every 24 hours; the third group will be assigned the device containing Beclomethasone/ Formoterol/ Glycopyrronium 100/6/12.5 mcg (Trimbow) with doses of two inhalations every 12 hours; the forth group will be assigned the device containing Budesonide/Formoterol/Glycopyrronium 160/4.8/7.2 mcg with doses of two inhalations every 12 hours. Each patient will be given a 100 μg salbutamol device as rescue medication.

Once the study medication is assigned, they will be instructed in technique and dosage, and a corresponding dose will be applied. A blood sample will be taken for a blood count and IgE test and Th2 and Th17 inflammatory profile cytokines. After 30 minutes of application of the study medication, impulse oscillometry, slow spirometry and forced spirometry will be performed. After 2 hours of application of study medication, impulse oscillometry, slow spirometry and forced spirometry will be performed. After 4 hours of application of study medication, impulse oscillometry, slow spirometry and forced spirometry will be performed. At the end of the respiratory function tests, the patient will be referred to the imaging service for tomography evaluation if it is not available with volumetry in the last year. Adverse events will be measured at baseline, for the safety outcome. The patient will be instructed in the use of the assigned medication, technique, frequency of use, as well as information and training on possible side effects. Visit 1 will be scheduled the next day without a window period.

Follow-up visit 1 (Visit 1, Day 1): Changes in respiratory symptoms, presence of adverse events, and use of concomitant medication will be questioned and documented. Symptom diary will be reviewed. It will be confirmed that the patient has not applied the morning dose of study medication. Dyspnea questionnaire (mMRC) and quality of life questionnaire (CAT) will be completed. Pulmonary function tests will be performed: FeNO, impulse oscillometry, slow spirometry, forced spirometry and simple plethysmography. Standard doses of SABA (400 mcg of salbutamol) will be applied and after 20 minutes post-bronchodilator tests of impulse oscillometry, slow spirometry and forced spirometry will be performed. The patient will be instructed in the technique of inhalation of study medication and a corresponding dose will be applied. Study medication will be provided for one month of treatment. A symptom diary will be provided and a follow-up visit 2 will be scheduled 30 days after the randomization visit.

Follow-up visit 2 (Visit 2, 30 days -2/+1 day): Exacerbations during the period, frequency of adverse events, newly diagnosed comorbidities and use of concomitant medication will be questioned and documented. Symptom diary will be reviewed. Devices dispensed at visit 1 will be reviewed to calculate adherence to treatment (≥80%). It will be confirmed that the patient has not applied the morning dose of study medication. Dyspnea questionnaire (mMRC), quality of life questionnaire (Saint George and CAT), and adherence to inhaled medication questionnaire (TAI) will be completed. Baseline pulmonary function tests will be performed: FeNO, impulse oscillometry, slow spirometry, forced spirometry and simple plethysmography. Short-acting bronchodilator (SABA) will be applied, the patient will be left to rest for 20 minutes. Post-bronchodilator tests will be initiated in the following order: impulse oscillometry, slow spirometry, forced spirometry. The patient will be instructed in the technique of inhalation of study medication and a corresponding dose will be applied. Study medication will be provided for two months of treatment. A symptom diary will be provided and a follow-up visit 3 will be scheduled 12 weeks after the randomization visit. Instructions for said visit will be given.

Follow-up visit 3 (Visit 3, 12 weeks -2/+1 day): Exacerbations during the period, frequency of adverse events, newly diagnosed comorbidities and use of concomitant medication will be questioned and documented. Symptom diary will be reviewed. Devices dispensed at visit 1 will be reviewed to calculate adherence to treatment (≥80%). It will be confirmed that the patient has not applied the morning dose of study medication. Dyspnea questionnaire (mMRC), quality of life questionnaire (Saint George and CAT), and adherence to inhaled medication questionnaire (TAI) will be completed. Baseline pulmonary function tests will be performed: FeNO, impulse oscillometry, slow spirometry, forced spirometry and simple plethysmography. Standard doses of SABA (400 mcg of salbutamol) will be applied and after 20 minutes post-bronchodilator tests of impulse oscillometry, slow spirometry and forced spirometry will be performed. Participation in the protocol will be terminated and monitoring by the NIRD Tobacco and COPD clinic will continue.

ELIGIBILITY:
Inclusion Criteria:

* Subject capable of understanding instructions and giving her consent for participation.
* Diagnosis of COPD or chronic bronchitis without obstruction due to biomass smoke exposure:

  1. Diagnosis of COPD according to GOLD guidelines 2023 with: >100 hours-year of biomass exposure index, and with a post-bronchodilator spirometry FEV1 > 70% of predicted value.
  2. Diagnosis of Chronic Bronchitis without obstruction with at least >100 hours-year of biomass smoke exposure index or more than 10 years of continued exposure to biomass smoke, and with 1) antecedent of chronic bronchitis, and 2) post-bronchodilator spirometry FEV1/FVC >0.7.
* Able to attend all visits.
* Cooperative patients with adequate understanding and skill in using inhalers, or with caregivers capable of administering medications and filling out a daily symptom diary.
* Stable patients, with no history of exacerbations in the last 4 weeks before inclusion.

Exclusion Criteria:

* Pregnancy or in the breastfeeding period.
* Documented allergy or intolerance to any of the study medications.
* History of clinically significant bronchiectasis, tuberculosis, recent respiratory infection (4 weeks), or cardiovascular comorbidity that contraindicates pulmonary function tests or that influences their status and functional class.
* Patients with suspicion or history of cancer.
* Uncontrolled diseases: acute hyperthyroidism, acute uncontrolled DM2, acid-peptic disease that causes bleeding, uncontrolled hematological diseases, etc. In general, any decompensated disease that, in the opinion of the principal investigator, may influence the results of the study.

Ages: 35 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Change in impulse oscillometry | 3 months
  To quantify the change in impulse oscillometry (post-bronchodilator) change in total resistance measured in percentage change from baseline change R5-R20 and/or AX for the patients who used Vilanterol / Umeclidinium 25/62.5 mcg once daily = ANORO®; Fluthicasone / Vilanterol / Umeclidinium 100/25/62.5 mcg once daily= TRELEGY®; Beclomethasone / Formoterol / Glycopyrronyum 100/6/12.5 mcg; two inhalations twice daily = TRIMBOW®; and Budesonide / Formoterol / Glycopyrronyum 160/4.8/7.2 mcg two inhalations twice daily= TRIXEO®.

SECONDARY OUTCOMES:
Change of resistences in impulse oscillometry | 30 minutes, 2 hours, 4 hours, 24 hours, 1 month, 3 months
  Quantify the change in R5, R20, R5-R20 [kPa/(L/s)]
Change of resistences in impulse oscillometry | 30 minutes, 2 hours, 4 hours, 24 hours, 1 month, 3 months
  Quantify the change in Ax [kPa/L]
Change of total resistances in pletismography | 30 minutes, 2 hours, 4 hours, 24 hours, 1 month, 3 months
  Change in total resistances (kPa*s/L), measured by plethysmography.
Chance in lung function in spirometry | 30 minutes, 2 hours, 4 hours, 24 hours, 1 month, 3 months
  Change in FEV1, and FVC, both in liters.
Chance in lung function in spirometry | 30 minutes, 2 hours, 4 hours, 24 hours, 1 month, 3 months
  Change in FEV1, and FVC, both percentage of predicted
Chance in FEF25-75 in spirometry | 30 minutes, 2 hours, 4 hours, 24 hours, 1 month, 3 months
  Change in FEF25-75 (L/s)
Chance in MMEF(L/s) in spirometry | 30 minutes, 2 hours, 4 hours, 24 hours, 1 month, 3 months
  Change in MMEF(L/s)
Adherence assesment | 3 months
  Quantify adherence to treatment according to the type of inhaler.
Change in Fractional exhaled nitric oxide | 3 months
  Change in exhaled fraction of nitric oxide measured by parts per billion.
Change in Chronic Obstructive Pulmonary Disease Assesment Test | 3 months
  Change in quality of life in Chronic Obstructive Pulmonary Disease Assesment Test score
Change in Saint George Respiratory Questionnaire | 3 months
  Change in quality of life in the Saint George respiratory questionnaire scores
Change in dypsnea by modified Medical Research Council score | 3 months
  Change in dyspnea score measured by the modified Medical Research Council test

CONTACTS AND LOCATIONS:
Locations (1):
- Insituto Nacional de Enfermedades Respiratorias "Ismael Cosío Villegas", Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: Yes
The data will be collected on the redCap platform and may be shared in Excel CSV format upon request after the results are published.
Supporting Information: Study Protocol, SAP
Time Frame: The IPD data will be available for sharing after the results are published. The data will me available for one year.
Access Criteria: The information may be requested by researchers who wish to carry out a meta-analysis. The main author will evaluate the applications for sharing the data.

REFERENCES:
- [Background] Perez-Padilla R, Regalado J, Vedal S, Pare P, Chapela R, Sansores R, Selman M. Exposure to biomass smoke and chronic airway disease in Mexican women. A case-control study. Am J Respir Crit Care Med. 1996 Sep;154(3 Pt 1):701-6. doi: 10.1164/ajrccm.154.3.8810608.
- [Background] Regalado J, Perez-Padilla R, Sansores R, Paramo Ramirez JI, Brauer M, Pare P, Vedal S. The effect of biomass burning on respiratory symptoms and lung function in rural Mexican women. Am J Respir Crit Care Med. 2006 Oct 15;174(8):901-5. doi: 10.1164/rccm.200503-479OC. Epub 2006 Jun 23. PMID 16799080
- [Background] García-Ochoa R, Rivera-Castañeda P, Bracamonte-Sierra Á. Desigualdad social en torno al uso de tecnologías energéticamente eficientes en México. El caso de la política de normalización de refrigeradores. Estudios Sociales; 29. Epub ahead of print 16 June 2019. DOI: 10.24836/es.v29153.722.
- [Background] Luo B, Niu .J Short-term effects of rural indoor air pollution on respiratory health and urine biomarkers of college students in the northwestern China. ISEE Conference Abstracts 2020; 2020: isee.2020.virtual.P-1226.
- [Background] GOLD. GLOBAL STRATEGY FOR PREVENTION, DIAGNOSIS AND MANAGEMENT OF COPD: 2023 Report, https://goldcopd.org/2023-gold-report-2/ (2023).
- [Background] Vestbo J, Lange P. Can GOLD Stage 0 provide information of prognostic value in chronic obstructive pulmonary disease? Am J Respir Crit Care Med. 2002 Aug 1;166(3):329-32. doi: 10.1164/rccm.2112048. PMID 12153965
- [Background] GBD 2016 Risk Factors Collaborators. Global, regional, and national comparative risk assessment of 84 behavioural, environmental and occupational, and metabolic risks or clusters of risks, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1345-1422. doi: 10.1016/S0140-6736(17)32366-8. PMID 28919119
- [Background] Anzueto A, Heijdra Y, Hurst RJ. Controversies ni COPD: ERS Monograph. European Respiratory Society, 2015.
- [Background] Ramirez-Venegas A, Sansores RH, Quintana-Carrillo RH, Velazquez-Uncal M, Hernandez-Zenteno RJ, Sanchez-Romero C, Velazquez-Montero A, Flores-Trujillo F. FEV1 decline in patients with chronic obstructive pulmonary disease associated with biomass exposure. Am J Respir Crit Care Med. 2014 Nov 1;190(9):996-1002. doi: 10.1164/rccm.201404-0720OC. PMID 25172140
- [Background] Ramirez-Venegas A, Torres-Duque CA, Guzman-Bouilloud NE, Gonzalez-Garcia M, Sansores RH. SMALLa AIRWAY DISEASE IN COPD ASSOCIATED TO BIOMASS EXPOSURE. Rev Invest Clin. 2019;71(1):70-78. doi: 10.24875/RIC.18002652. PMID 30810542
- [Background] Han MK, Agusti A, Celli BR, Criner GJ, Halpin DMG, Roche N, Papi A, Stockley RA, Wedzicha J, Vogelmeier CF. From GOLD 0 to Pre-COPD. Am J Respir Crit Care Med. 2021 Feb 15;203(4):414-423. doi: 10.1164/rccm.202008-3328PP. No abstract available. PMID 33211970
- [Background] Camp PG, Ramirez-Venegas A, Sansores RH, Alva LF, McDougall JE, Sin DD, Pare PD, Muller NL, Silva CI, Rojas CE, Coxson HO. COPD phenotypes in biomass smoke- versus tobacco smoke-exposed Mexican women. Eur Respir J. 2014 Mar;43(3):725-34. doi: 10.1183/09031936.00206112. Epub 2013 Oct 10. PMID 24114962
- [Background] Ramírez-Venagas A. Efficacy and Safety of ICS/LABA vs. LAMA/LABA in Patients With Different COPD Phenotypes. NCT05342558, https://classic.clinicaltrials.gov/ct2/show/NCT05342558 (2022).
- [Background] Han MK, Ye W, Wang D, White E, Arjomandi M, Barjaktarevic IZ, Brown SA, Buhr RG, Comellas AP, Cooper CB, Criner GJ, Dransfield MT, Drescher F, Folz RJ, Hansel NN, Kalhan R, Kaner RJ, Kanner RE, Krishnan JA, Lazarus SC, Maddipati V, Martinez FJ, Mathews A, Meldrum C, McEvoy C, Nyunoya T, Rogers L, Stringer WW, Wendt CH, Wise RA, Wisniewski SR, Sciurba FC, Woodruff PG; RETHINC Study Group. Bronchodilators in Tobacco-Exposed Persons with Symptoms and Preserved Lung Function. N Engl J Med. 2022 Sep 29;387(13):1173-1184. doi: 10.1056/NEJMoa2204752. Epub 2022 Sep 4. PMID 36066078
- [Background] Borrill ZL, Houghton CM, Woodcock AA, Vestbo J, Singh D. Measuring bronchodilation in COPD clinical trials. Br J Clin Pharmacol. 2005 Apr;59(4):379-84. doi: 10.1111/j.1365-2125.2004.02261.x. PMID 15801931
- [Background] Manoharan A, Morrison AE, Lipworth BJ. Effects of Adding Tiotropium or Aclidinium as Triple Therapy Using Impulse Oscillometry in COPD. Lung. 2016 Apr;194(2):259-66. doi: 10.1007/s00408-015-9839-y. Epub 2016 Jan 13. PMID 26758884
- [Background] Sana A, Somda SMA, Meda N, Bouland C. Chronic obstructive pulmonary disease associated with biomass fuel use in women: a systematic review and meta-analysis. BMJ Open Respir Res. 2018 Jan 12;5(1):e000246. doi: 10.1136/bmjresp-2017-000246. eCollection 2018. PMID 29387422
- [Background] Ramirez-Venegas A, Velazquez-Uncal M, Perez-Hernandez R, Guzman-Bouilloud NE, Falfan-Valencia R, Mayar-Maya ME, Aranda-Chavez A, Sansores RH. Prevalence of COPD and respiratory symptoms associated with biomass smoke exposure in a suburban area. Int J Chron Obstruct Pulmon Dis. 2018 May 25;13:1727-1734. doi: 10.2147/COPD.S156409. eCollection 2018. PMID 29872290
- [Background] Orduz García CE, Toro MV, Gómez JC. EPOC, BRONQUITIS CRÓNICA YSÍNTOMAS RESPIRATORIOS, ASOCIADOS ALA CONTAMINACIÓN POR PM10 EN LA CIUDAD DE MEDELLÍN (COLOMBIA). Revista Med 2013; 21: 21-28.
- [Background] Rivera RM, Cosio MG, Ghezzo H, Salazar M, Perez-Padilla R. Comparison of lung morphology in COPD secondary to cigarette and biomass smoke. Int J Tuberc Lung Dis. 2008 Aug;12(8):972-7. PMID 18647460
- [Background] Graham BL, Steenbruggen I, Miller MR, Barjaktarevic IZ, Cooper BG, Hall GL, Hallstrand TS, Kaminsky DA, McCarthy K, McCormack MC, Oropez CE, Rosenfeld M, Stanojevic S, Swanney MP, Thompson BR. Standardization of Spirometry 2019 Update. An Official American Thoracic Society and European Respiratory Society Technical Statement. Am J Respir Crit Care Med. 2019 Oct 15;200(8):e70-e88. doi: 10.1164/rccm.201908-1590ST. PMID 31613151
- [Background] Stanojevic S, Kaminsky DA, Miller MR, Thompson B, Aliverti A, Barjaktarevic I, Cooper BG, Culver B, Derom E, Hall GL, Hallstrand TS, Leuppi JD, MacIntyre N, McCormack M, Rosenfeld M, Swenson ER. ERS/ATS technical standard on interpretive strategies for routine lung function tests. Eur Respir J. 2022 Jul 13;60(1):2101499. doi: 10.1183/13993003.01499-2021. Print 2022 Jul. PMID 34949706

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-13): https://cdn.clinicaltrials.gov/large-docs/42/NCT06571942/Prot_SAP_000.pdf